CLINICAL TRIAL: NCT07132255
Title: Platform Construction and Clinical Application of 5G Technology for Remote Operation of the R-One™ Robot in Percutaneous Coronary Intervention
Brief Title: The Efficacy and Safety Evaluation of 5G Tele-PCI Using R-OneTM
Acronym: tele-PCI
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Cathbot (Shanghai) Robot Co., Ltd (Industry)
Collaborators: People's Hospital of Xinjiang Uygur Autonomous Region (Other); Karamay Central Hospital of Xinjiang (Unknown); The First Hospital of Kashgar Prefecture (Unknown); Jimusar People's Hospital (Unknown); Luopu People's Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-One-20241121231; 20241121231 (Other Grant/Funding Number: Science And Technology Department Of Xinjiang Uygur Autonomous Region)
Record Dates: First submitted 2025-08-11; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Coronary Artery Disease (CAD); Percutaneous Coronary Intervention (PCI)
Keywords: PCI; tele-PCI; CAD
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: This prospective multicenter exploratory clinical study is conducted simultaneously at one remote control center and four on-site operative centers. 60 eligible subjects are randomly allocated into either on-site R-One-assisted PCI group or R-One-assisted tele-PCI group. The surgical team will perform robot-assisted PCI procedures while researchers systematically document device performance metrics to evaluate the remote operational performance of R-One.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- R-One assisted tele-PCI (Experimental): The investigational device was R-One Vascular Interventional Navigation Control System developed and produced by Robocath, and was composed of a platform (instruction unit, robot, support joint arm), a consumable set (cartridge, instruction unit protective sleeve), and a remote workstation.
  To achieve remote surgery, remote communication workstations need to be configured at all locations where remote surgery is performed.
  The remote communication workstation of local operating room will establish the virtual surgery, and the remote communication workstation of the remote control side needs to join the virtual surgery through the invitation code to establish remote control between the two places.
  After the virtual surgery is established, the two communication workstations need to incorporate the robots nearby into the operation. In this way, the two control consoles can achieve remote control and data exchange.
  Interventions: Device: R-One assisted tele-PCI
- R-One assisted on-site PCI (Active Comparator): The product is designed with a master-slave control, which inserts and retracts guidewires, balloons and stent catheters via a remote-controlled robotic arm. The surgeon inputs the movements through the handle at the master end, and the robot replicates the surgeon's hand movements from the slave end to complete the surgical operation.
  Interventions: Device: R-One assisted on-site PCI

INTERVENTIONS:
Device: R-One assisted tele-PCI — Surgeons perform operations using R-One vascular interventional navigation control system from remote control center via 5G. robotic slave executes at procedure site.
  Arms: R-One assisted tele-PCI
Device: R-One assisted on-site PCI — Surgeons perform operations by controlling robot from local console .
  Arms: R-One assisted on-site PCI

SUMMARY:
Patients with coronary artery disease requiring PCI treatment were enrolled in the study.

All patients underwent PCI with the robotic R-OneTM System (R-One Vascular Robotics, Cathbot). The system was designed for coronary PCI and consists of 2 major components: the command unit and a bedside robot. The command unit is a radiation-shielded, mobile workstation that was positioned in the corner of the catheterization laboratory. The interventional cardiologist sits at the command unit and remotely performs the PCI using the console joysticks. Commands from the control console are delivered as electrical signals along a communication cable that runs from the control console to the robotic drive, on which a sterile cassette is placed. The cassette, which is loaded with the robot and connected to the guiding catheters, imposes axial and rotational forces on the intracoronary devices. Fluoro-scopic, electrocardiographic, and hemodynamic images are "slaved" to the duplicate monitors inside the cockpit, enabling visualization from a closer distance.

After completion of diagnostic angiography, the guiding catheter was positioned at the ostium of the coronary artery and connected to the disposable cassette on the robotic drive. The guidewire was loaded into the cassette before starting the robotic-enhanced PCI. The treatment plan is decided by the doctor according to the patients' situation. All intracoronary devices were to be manipulated exclusively by the robotic system, with bailout to manual conversion when needed.

The primary endpoints were clinical procedural success and device technical success. The necessary sample size for testing the endpoint of clinical and technical procedural success was calculated on the basis of the target value. The statistical analysis results show that the lower limit of the 95% confidence interval of the clinical success rate and the technical success rate of the operation is greater than 90% of the target value, and the invalid hypothesis is rejected. Both primary endpoints had to be met for the study to be declared successful. Data were analyzed on an intention-to-treat basis. Standard summary statistics were calculated for all patient and study outcome variables. Continuous variables were summarized using estimated means, standard deviations, minimums, maximums, medians, and interquartile ranges. Categorical data were summarized using frequencies, percentages, and 95% confidence interval.

DETAILED DESCRIPTION:
1. Purpose To evaluate the effectiveness and safety of 5G-enabled remote control of the R-OneTM vascular interventional navigation control system for percutaneous coronary interventions.
2. Research design A prospective, multicenter, exploratory clinical trial. Subjects who met the inclusion criteria and did not meet the exclusion criteria were enrolled into the clinical study, and the subjects are randomly grouped by using the interactive web response system (IWRS) applet (MedLand Centralized Randomization Management System). The surgeons completed the robotic-assisted surgical operation using the investigational device during cardiovascular PCI treatment. The investigator is also required to evaluate the performance of the investigational device during the procedure and ultimately determine the safety and efficacy of its clinical application.
3. Device The investigational device was R-One Vascular Interventional Navigation Control System developed and produced by Robocath, and was composed of a platform (instruction unit, robot, support joint arm), a consumable set (cartridge, instruction unit protective sleeve), and a remote workstation.
4. Scope of Trial The subjects scope of the clinical trial: Patients requiring cardiovascular PCI.
5. Experimental Procedure Information of all the patients who have signed the Informed Consent Form and actually pass the screening will be registered in the screening/enrollment log sheet. If a subject is excluded from the trial, the investigator should specify the reasons for screening failure. If a subject is enrolled in the trial but does not use the investigational device, the reason should also be recorded.

All subjects enrolled in the trial will be given a corresponding enrollment number.

72-hour pre-operative collected ECG, cardiac enzyme, and concomitant medication records.

Operation day visit The investigator is also required to complete the cardiology robot-assisted surgical treatment using the investigational device and record the procedure, LED Scale, SME Scale, and device Performance Evaluation Pre-discharge visit The investigator shall collect the blood test, creatinine, ECG. cardiac enzyme, concomitant medication records.

1 month post-operative visit The investigator shall collect the concomitant medication records.

Application method of the investigational device Subjects who meet the inclusion criteria and do not meet the exclusion criteria will be enrolled in the clinical study and the surgeon will complete the therapeutic treatment on the subject while performing the cardiology PCI procedure.

The investigational devices should be used by investigators respectively during the surgical treatment according to product instructions. Surgeons who would participate in the trial and use the study device should have completed at least 80 PCI procedures and need to be trained and supervised by the physician who completed the animal experiments using the investigational device.

General procedure of a surgical operation

Connect the power cord to the mains.

1. Connect the power cord to the mains.
2. Load the instruction unit, ensuring that the positioning mark on the base and that on the radiation-proof screen overlap.
3. Switch on the system
4. Activate the system.
5. Prepare R-One consumables kit.
6. Install the instruction unit protective sleeve.
7. Install the cartridge.
8. Install the robot.
9. Attach the Y-connector clip to the cartridge.
10. Insert the guide wire in the cartridge.
11. Navigate the guide wire through the instruction unit
12. Move the control lever and actuate the guidewire
13. Fix the guidewire
14. Insert the catheter into the cartridge
15. Navigate the catheter through the instruction unit
16. Move the control lever and actuate the catheter
17. Securing catheter
18. Simultaneous navigate the guidewire and catheter from the instruction unit
19. Place the guide wire in the alternate path as a backup
20. Place the catheter in the alternate path as a backup
21. Adjust the robot position

6. Primary Evaluation Indicators

1. Clinical success rate of the surgery

   Calculation formula:

   Clinical success rate = number of subjects that were clinical successes ÷ number of subjects that received surgical treatment × 100%.

   Evaluation Method:

   Clinical surgical success

   Definition of clinical surgical success:

   The target lesion was treated with test device, and the residual stenosis in the target vessel (visual description by angiography) reduced to less than 30% after PCI and a thrombolysis in myocardial infarction (TIMI) grade of 3.

   No major adverse cardiovascular events (MACE) occurred in the hospital.
2. Success rate of surgical techniques

Calculation formula:

Technical success rate = number of subjects that were technical successes ÷ number of subjects received surgical treatment × 100%

Evaluation Method:

Technical success of the surgery

Definition of technical success:

The Robot-assisted PCI procedure was successfully completed without any unplanned manual assistance or shift to manual operation.

Definition of planned manual assistance:

During robotic surgery: Reposition of guidewires or stents/balloons, manual translation/rotation of guidewires or stents/balloons to guiding catheters, reposition of guiding catheters and usage of any device that is not compatible with the robotic platform

Definition of unplanned manual assistance:

Manual translation/rotation of the guidewire and/or manual translation of the stent/balloon once the guidewire has left the guiding catheter

Definition of the shift to manual operation:

Any situation during the PCI procedure that results in the shift to manual operation.

System restart failure during robotic surgery.

7. Secondary Evaluation Indicators

1. Procedure duration

   Calculation formula:

   Procedure duration = arterial sheath removal time - arterial sheath insertion time.
2. Duration of robot-assisted treatment

   Calculation formula:

   Robot-assisted treatment duration = time when the robot finish moving the guidewire away from the coronary vessel - time when the robot starts manipulating the guidewire.
3. Radiation exposure to the patient Evaluation Method: Measure and record dose exposure by angiography (DSA)
4. Radiation exposure to surgeons Evaluation Method: Detect radiation through radiation dosimeters. Two dosimeters will be used simultaneously during the procedure. One is placed on the operating table and the other is worn by the surgeon to measure the radiation dose exposed to the surgeon. Both dosimeters will be calibrated once a day before use and reset to zero before each PCI procedure. Radiation readings from the dosimeter will be recorded when the first guidewire is inserted into the vessel and the last guidewire is pulled out of the vessel.
5. Contrast dose Evaluation Method: Record the contrast dose used during intra-operative angiography
6. MACE Evaluation Method: Record the MACE in-hospital and within 1 month (30±7 days) after the PCI procedure
7. Product performance indicators Evaluation of intraoperative physiological load of surgeons. Evaluation Method: Surgeons are required to complete the Local Experienced Discomfort Questionnaire (LED scale) in time after the surgery in order to provide a retrospective evaluation of the physiological sensations during the procedure in the way of visual analog scale.
8. Intraoperative psychological load evaluation of surgeons Evaluation Method: Surgeons are required to complete the Subjective Mental Effort Questionnaire (SME scale) in time after the surgery in order to provide a retrospective evaluation of the mental feelings during the procedure in the way of visual analog scale.
9. Intraoperative remote control performance evaluation of surgeons Evaluation Method: Both remote and local surgeons are required to promptly complete postoperative subjective assessments of intraoperative operational experience, including real-time responsiveness of remote surgical maneuvers, image quality of remote high-definition DSA (Digital Subtraction Angiography) imaging, transmission immediacy of remote DSA images, immediacy and stability of remote audio transmission, and operational flexibility of the slave-side bedside manipulator arms.
10. Incidence rate of serious system malfunction Calculation formula: Incidence rate of serious system malfunction = Number of procedures with serious system malfunction during robot-assisted surgery ÷ Number of procedures in which robot-assisted surgery was performed × 100%.

    Definition of serious system malfunction Evaluation Method: System malfunctions that occur during robot-assisted surgery that are difficult to repair in a short period of time and can have a serious impact on the surgical process or options.
11. The occurrences of repairable system malfunction Evaluation Method: Definition of repairable system malfunction: Simple malfunctions that occur during robot-assisted surgery that can be repaired by a technician or the surgical team and do not have a serious impact on the surgical process or options.
12. Evaluation of Device Usability Evaluation Method: Record the performance of the investigational device from preoperative preparation to the end of the procedure. Investigators are required to complete the Device Performance Evaluation Form after surgery and provide a retrospectively evaluation of performance of the investigational device during the trial.
13. Indicators for Safety Evaluation Subjects' laboratory test results collected during the screening period, operation day, pre-discharge and 1-month post-operative visit, and information of adverse events during the clinical trial, as well as investigational device-related adverse events and serious adverse events.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age ≤ age ≤ 80 years of age.
* Have clinical indication(s) for PCI and need to be treated with a PCI procedure.
* Subjects voluntarily signed an informed consent form and were willing to complete follow-up visits.
* Visual description of target lesion diameter stenosis ≥70% (or ≥50% accompanied with clinical evidence of myocardial ischemia within that range;
* 2.5 mm ≤reference vessel diameter by visual description ≤ 4.0 mm.
* Target lesion length ≤34.0 mm by visual description (If it is made up of multiple small lesions, the distance of which should not exceed 10 mm) and can be fully covered by a single stent. There are no less than 2.0 mm normal segmental vessels at the proximal and distal margins of the diseased region.
* ≤2 target vessels to be treated, one single stent for each target lesion per target vessel, and target lesions can not be treated through stages.

Exclusion Criteria:

* Subjects have undergone other PCI within 72 hours prior to the R-One PCI procedure;
* Subjects have undergone PCI within 30 days prior to the R-One PCI procedure and have experienced a MACE or other serious adverse event;
* Acute myocardial infarction (MI) within one week prior to scheduled R-One PCI procedure;
* Severe heart failure (NYHA ≥ Class III);
* Cardiogenic shock within 48 hours prior to the PCI procedure;
* Pregnant and lactating women, or women with plans to become pregnant during the clinical trial;
* Subjects with allergies to aspirin, heparin, clopidogrel, contrast media, metallic materials and rapamycin;
* Subjects with a platelet count <100 x 109/L or >700 x 109/L and a white blood cell (WBC) count <3 x 109/L (e.g., thrombocytopenia, thrombocytosis, neutropenia or leukopenia);
* Subjects with creatinine levels ≥ 177 umol/L;
* Subjects had a stroke within 30 days prior to the planned R-One PCI procedure.
* Subjects with an active peptic ulcer or upper gastrointestinal hemorrhage within 6 months prior to the PCI procedure.
* Subjects with a history of massive haemorrhage or coagulation disorder, or refusal of blood transfusion within the previous 6 months.
* Subjects are currently enrolled in another clinical study that has not yet completed the entire follow-up period.
* The investigators determined that the patient was not applicable for robot-assisted PCI.
* TIMI blood flow grade of <3 for the target lesion.
* In-stent restenosis, or the target vessel has implanted a stent previous which in close proximity to the target lesion.
* Need other treatments (e.g., atherectomy or laser treatment) in addition to balloon angioplasty and stentoplasty.
* Coronary anatomy deemed unsuitable for robot-assisted PCI as determined by the operator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-14 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Clinical success rate of the surgery | Operation day
  Calculation formula:
  Clinical success rate = number of subjects that were clinical successes ÷ number of subjects that received surgical treatment × 100%.
  Evaluation method:
  The target lesion was treated with test device, and the residual stenosis in the target vessel (visual description by angiography) reduced to less than 30% after PCI and a TIMI grade of 3.
  No major adverse cardiovascular events (MACE) occurred in the hospital.
Success rate of surgical techniques | Operation day
  Calculation formula:
  Technical success rate = number of subjects that were technical successes ÷ number of subjects received surgical treatment × 100%
  Evaluation method:
  The Robot-assisted PCI procedure was successfully completed without any unplanned manual assistance or shift to manual operation.
  Definition of planned manual assistance:
  During robotic surgery: Reposition of guidewires or stents/balloons, manual translation/rotation of guidewires or stents/balloons to guiding catheters, reposition of guiding catheters and usage of any device that is not compatible with the robotic platform
  Definition of unplanned manual assistance:
  Manual translation/rotation of the guidewire and/or manual translation of the stent/balloon once the guidewire has left the guiding catheter
  Definition of the shift to manual operation:
  Any situation during the PCI procedure that results in the shift to manual operation.
  System restart failure during robotic surgery

SECONDARY OUTCOMES:
Procedure duration | Operation day
  Procedure duration = arterial sheath removal time - arterial sheath insertion time
Duration of robot-assisted treatment | Operation day
  Robot-assisted treatment duration = time when the robot finish moving the guidewire away from the coronary vessel - time when the robot start to move the guidewire away from the guiding catheter
Radiation exposure to the patient | Operation day
  Evaluation Method: Measure and record dose exposure by angiography (DSA)
Radiation exposure to surgeons | Operation day
  Detect radiation through radiation dosimeters. Two dosimeters will be used simultaneously during the procedure. One is placed on the operating table and the other is worn by the surgeon to measure the radiation dose exposed to the surgeon. Both dosimeters will be calibrated once a day before use and reset to zero before each PCI procedure. Radiation readings from the dosimeter will be recorded when the first guidewire is inserted into the vessel and the last guidewire is pulled out of the vessel.
Contrast dose | Operation day
  Record the contrast dose used during intra-operative angiography
MACE | Operation day and 1 month post-operative
  Record the in-hospital MACE of subjects Record the MACE occurred 1 month (30±7 days) after the PCI procedure

OTHER OUTCOMES:
Intraoperative physiological load evaluation of surgeons | Operation day
  Surgeons are required to complete the Local Experienced Discomfort Questionnaire (LED scale) in time after the surgery in order to provide a retrospective evaluation of the physiological sensations during the procedure in the way of visual analog scale.0 = No discomfort at all, and 10 = Very uncomfortable.
Intraoperative psychological load evaluation of surgeons | Operation day
  Surgeons are required to complete the Subjective Mental Effort Questionnaire (SME scale) in time after the surgery in order to provide a retrospective evaluation of the mental feelings during the procedure in the way of visual analog scale. 0 = Not difficult at all, and 100 = Extremely difficult.
Intraoperative Remote Control Performance Evaluation of surgeons | Operation day
  Calculation formula:
  Incidence rate of serious system malfunction = Number of procedures with serious system malfunction during robot-assisted surgery ÷ Number of procedures in which robot-assisted surgery was performed × 100%.
  Evaluation Method:
  Definition of serious system malfunction: System malfunctions that occur during robot-assisted surgery that are difficult to repair in a short period of time and can have a serious impact on the surgical process or options.
The occurrences of repairable system malfunction | Operation day
  Definition of repairable system malfunction: Simple malfunctions that occur during robot-assisted surgery that can be repaired by a technician or the surgical team and do not have a serious impact on the surgical process or options.
Evaluation of Device Usability | Operation day
  Record the performance of the investigational device from preoperative preparation to the end of the procedure.
  Investigators are required to complete the Device Performance Evaluation Form after surgery and provide a retrospectively evaluation of performance of the investigational device during the trial.
Indicators for Safety Evaluation | 72 hours pre, operation day, pre-discharge and 1-month post-operative
  Subjects' laboratory test results collected during the screening period, operation day, pre-discharge and 1-month post-operative visit, and information of adverse events during the clinical trial, as well as investigational device-related adverse events and serious adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Yining Yang, Principal Investigator — People's Hospital of Xinjiang Uygur Autonomous Region
Locations (5):
- China (5):
  - Jimsar People's Hospital, Jimsar, Xinjiang Uygur Autonomous Region
  - Karamay Central Hospital of Xinjiang, Karamay, Xinjiang Uygur Autonomous Region
  - The First Hospital of Kashgar Prefecture, Kashgar, Xinjiang Uygur Autonomous Region
  - Luopu People's Hospital, Luopu, Xinjiang Uygur Autonomous Region
  - People's Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang Uygur Autonomous Region

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol (2025-03-01): https://cdn.clinicaltrials.gov/large-docs/55/NCT07132255/Prot_000.pdf
  • Statistical Analysis Plan (2025-03-01): https://cdn.clinicaltrials.gov/large-docs/55/NCT07132255/SAP_001.pdf
  • Informed Consent Form (2025-03-01): https://cdn.clinicaltrials.gov/large-docs/55/NCT07132255/ICF_002.pdf